CLINICAL TRIAL: NCT07332325
Title: STeroids and Enhanced Spectrum Antibiotics for the Treatment of Patients in Africa With Refractory Sepsis (STARS Trial)
Brief Title: STeroids and Enhanced Spectrum Antibiotics for the Treatment of Patients in Africa With Refractory Sepsis
Acronym: STARS
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Scott Heysell, MD, Professor of Medicine, University of Virginia
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: HSR302304; 1U01AI192033-01 (NIH)
Record Dates: First submitted 2026-01-06; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Sepsis; Tuberculosis
Keywords: Sepsis; HIV; tuberculosis; Africa
MeSH Terms: conditions — Sepsis; Tuberculosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- No hydrocortisone/standard antimicrobial therapy (No Intervention): Standard of care
- Hydrocortisone/standard antimicrobial therapy (Experimental)
  Interventions: Drug: Hydrocortisone administration
- No hydrocortisone/enhanced spectrum antimicrobial therapy (Experimental)
  Interventions: Drug: Expanded antimicrobial therapy
- Hydrocortisone/enhanced spectrum antimicrobial therapy (Experimental)
  Interventions: Drug: Hydrocortisone administration; Drug: Expanded antimicrobial therapy

INTERVENTIONS:
Drug: Hydrocortisone administration — Immediate hydrocortisone at 200 mg IV daily for 7 days and a tapering schedule for an additional 7 days
  Arms: Hydrocortisone/enhanced spectrum antimicrobial therapy; Hydrocortisone/standard antimicrobial therapy
Drug: Expanded antimicrobial therapy — empiric initiation of the enhanced spectrum antimicrobial therapy regimen (rifampin, isoniazid, linezolid, and levofloxacin) for 14 days plus standard care which includes ceftriaxone for 7 days or diagnosis dependent conventional anti-TB therapy
  Arms: Hydrocortisone/enhanced spectrum antimicrobial therapy; No hydrocortisone/enhanced spectrum antimicrobial therapy

SUMMARY:
Sepsis, a life-threatening condition due to a dysregulated response to infection, is the leading cause of global mortality and is frequently driven by tuberculosis (TB) and drug-resistant bacteria in sub-Saharan Africa, particularly among people living with HIV. The current standard of care in the region, ceftriaxone, is insufficient as it does not address TB, drug-resistant bacteria, or adrenal insufficiency, which is common in HIV-related sepsis. Therefore, the investigators propose a randomized 2x2 factorial clinical trial to compare 28-day survival from sepsis between study participants who along with the standard of care receive 1) hydrocortisone to treat septic shock and 2) rifampin, isoniazid, levofloxacin and linezolid to treat TB and other drug-resistant bacteria in order to deliver important and scalable knowledge that may alter the standard of care for sepsis in HIV endemic settings of sub-Saharan Africa. Improving understanding of the physiology and treatment alternatives for HIV related critical illness globally will have reciprocal benefit for health in the U.S.

DETAILED DESCRIPTION:
Sepsis is defined as life-threatening organ dysfunction due to a dysregulated host response to infection and is the leading cause of global mortality. The World Health Organization has declared sepsis a global priority. Yet, little is known about sepsis in the global South and specifically sub-Saharan Africa where there are an estimated 17 million cases and 3.5 million attributable deaths per year. The majority of these patients are living with human immunodeficiency virus (HIV). The investigators have determined the leading cause of sepsis in this region is tuberculosis (TB) which is responsible for 25-30% of bloodstream infections in septic patients. TB sepsis is associated with 20-50% mortality rates with the majority of deaths occurring within the first 4-5 days of admission. Other causative pathogens include bacteria commonly or intrinsically resistant to third-generation cephalosporins which are the standard antimicrobial treatment for sepsis adopted from the global North. The investigators have also studied anti-TB pharmacokinetics/pharmacodynamics in septic patients and discovered considerably low circulating drug concentrations that are suboptimal for microbial kill. Concurrently, the investigators have also found a high burden of corticosteroid insufficiency in people with critical illness at collaborative study sites in Uganda and Tanzania. HIV and TB, independently and in combination, contribute to adrenal infection and endogenous steroid insufficiency. In further observational study, adults with sepsis at the collaborative study sites treated with corticosteroids have significantly improved survival from septic shock in-line with some, but not all, trials of adjunctive steroids in infection associated critical illness. Therefore, hypotheses are that immediate hydrocortisone administered over 7 days followed by a 7-day taper will improve 28 day mortality compared to the standard of care where corticosteroids are not administered, and that an enhanced antimicrobial regimen for 14 days to target TB and other drug-resistant bacteria of sepsis (rifampin, isoniazid, levofloxacin and linezolid) will improve 28 day mortality compared to the standard of care of ceftriaxone alone. These hypotheses will be tested through a randomized 2x2 factorial clinical trial where participants hospitalized with HIV and sepsis will be randomized to 1) hydrocortisone or the standard care without hydrocortisone, and 2) the enhanced antimicrobial regimen plus ceftriaxone or the standard care with ceftriaxone alone. This randomized 2x2 factorial clinical trial is strongly endorsed by Tanzanian and Ugandan stakeholders, utilizes drugs that are available within national formularies and regional pharmacies, and if successful will be scalable for adults with sepsis in HIV endemic regions of sub-Saharan Africa. Improved understanding of the physiology and treatment alternatives for HIV related critical illness globally will have reciprocal benefit for health in the U.S.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Male or female aged ≥18 years living with HIV
4. Admitted to hospital with 1) clinical concern for infection; 2) ≥2 qSOFA score criteria (Glasgow Coma Scale score <15, a respiratory rate ≥22, or a systolic blood pressure ≤90 mmHg or a mean arterial pressure of ≤65 mmHg)
5. Resident within a pre-defined geographic area to ensure TB clinic follow-up
6. For females of reproductive potential: use of highly effective contraception through 28 days

Exclusion Criteria:

1. Known active TB or receiving anti-TB therapy
2. Pregnancy or lactation. Women will undergo urine pregnancy screening. Pregnant people will be excluded due to lack of pharmacokinetic data for the expanded antibiotic regimen in pregnancy.
3. Known allergic reactions to the components of the interventional therapy
4. Treatment with another investigational drug or other intervention within one month
5. Known liver disease
6. Alcohol use > 14 standardized drinks per week and/or > 4 drinks per day for men and >7 standardized drinks per week and/or >3 drinks per day for women, defined as 14 grams of ethanol, as found in example 5 ounces of wine, 12 ounces of beer, or 1.5 ounces of 80 proof spirits
7. Positive serum cryptococcal antigen test
8. Current treatment with a drug known to have significant, non-correctable interaction with anti-TB therapy
9. Already receiving corticosteroids at the time of presentation to the hospital

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 344 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2029-03 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
Mortality | 28 days from date of randomization
  Primary outcome measure

SECONDARY OUTCOMES:
In-hospital mortality | from enrollment through hospitalization, an average of 14 days
  Mortality
6-month mortality | From the date of randomization until death or 180 days from randomization
  Mortality
Time to death | From date of randomization to death or 180 days from randomization
  Mortality
Incidence of new post-admission shock | From the time of enrollment through hospital discharge, an average of 14 days
  New post-admission shock
Duration of hospitalization | From the time of randomization until date of hospital discharge up to 180 days, or death if before hospital discharge
  Duration of hospitalization
Volume of IV fluids received | From the date of randomization until date of hospital discharge up to 180 days, or date of death if occurring before discharge
  Volume of IV fluids received
Adverse drug events during the 28-day study period | From date of randomization to 28 days post randomization or date of death if death occurred before 28 days
  Adverse drug events
Time to ambulation | From date of randomization until the date of first documented ambulation during hospitalization, or date of death from any cause, whichever came first, on average over 14 days, but up to 180 days
  Time to ambulation
Time to temperature normalization | From date of randomization until the date of first documented normal temperature during hospitalization, or date of death from any cause, whichever came first, on average over 14 days, but up to 180 days
  Time to temperature normalization
Lactate/delta lactate | From the date of randomization until the date of hospital discharge or the date of death if death occurred before discharge, on average 14 days
  Lactate concentration change
Capillary fill time/delta capillary fill time | From the date of randomization until the date of hospital discharge or the date of death if death occurred before discharge, on average 14 days
  Change in capillary fill time
Universal Vital Assessment score and delta Universal Vital Assessment score: component number one, heart rate | From the time of randomization to 72 hours after randomization
  Calculation of initial Universal Vital Assessment mortality risk score at randomization and 72 hours after randomization: component number one, measure heart rate
Universal Vital Assessment mortality risk score at randomization and 72 hours after randomization: component number two, respiratory rate | From time to randomization to 72 hours
  Calculation of initial Universal Vital Assessment mortality risk score at randomization and 72 hours after randomization: component number two, measure respiratory rate
Calculation of initial Universal Vital Assessment mortality risk score at randomization and 72 hours after randomization: component number three, systolic blood pressure | From time to randomization to 72 hours
  Calculation of initial Universal Vital Assessment mortality risk score at randomization and 72 hours after randomization: component number three, measure systolic blood pressure
Calculation of initial Universal Vital Assessment mortality risk score at randomization and 72 hours after randomization: component number four, oxygen saturation | From time to randomization to 72 hours
  Calculation of initial Universal Vital Assessment mortality risk score at randomization and 72 hours after randomization: component number four, measure oxygen saturation
Calculation of initial Universal Vital Assessment mortality risk score at randomization and 72 hours after randomization: component number five, glascow coma scale | From time to randomization to 72 hours
  Calculation of initial Universal Vital Assessment mortality risk score at randomization and 72 hours after randomization: component number five, record record level of consciousness by glascow come scale

CONTACTS AND LOCATIONS:
Overall Officials: Scott K Heysell, MD, MPH, Principal Investigator — University of Virginia; Christopher C Moore, MD, Principal Investigator — University of Virginia
Locations (4):
- Tanzania (2):
  - Sekou Toure Regional Referral Hospital, Mwanza
  - Kibong'oto Infectious Diseases Hospital, Sanya Juu
- Uganda (2):
  - Fort Portal Regional Referral Hospital, Fort Portal
  - Mbarara Regional Referral Hospital, Mbarara

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: Within one year of trial completion